CLINICAL TRIAL: NCT01232621
Title: A Randomized Pilot Study of Different Methods of Approaching Substitute Decision Makers Regarding Research Participation in the Intensive Care Unit: The Approach Study
Brief Title: The Approach Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-278
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Critical Care Trial Participation Consent by SDM
MeSH Terms: interventions — Consent Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician introduction (Experimental): Physicians will introduce Research Coordinators (RCs) by name to SDMs and acknowledge patient eligibility to participate in a study using a standardized script.
  Interventions: Other: Physician Introduction of research personnel
- Non-physician introduction (usual approach) (Active Comparator): RCs will either introduce themselves or be introduced by a non-physician member of the health care team.
  Interventions: Other: Physician Introduction of research personnel

INTERVENTIONS:
Other: Physician Introduction of research personnel — Physicians will introduce Research Coordinators (RCs) by name and acknowledge patient eligibility to participate in a research study using a standardized script.
  Other Names: Approach to Consent; Consent; Substitute Decision Maker

SUMMARY:
In the Approach Study, the investigators will study the 'process' by which Substitute Decision Makers (SDMs) are approached for consent for their loved one's participation in critical care research. The investigators will randomize SDMs of critically ill patients who are eligible to participate in any research study in operation to either 'physician introduction' of the research team or 'non-physician approach (non-physician)' in which research coordinators are introduced by allied health care team members or introduce themselves directly to SDMs. This study seeks to identify important features of the 'consent to research' process that can be modified to enhance both SDM satisfaction with the consent process and recruitment into critical care research studies.

DETAILED DESCRIPTION:
Rationale: Conduct of clinical research in the intensive care unit (ICU) presents challenges including the necessity to obtain consent for patients lacking decision-making capacity, operationalize research protocols under emergency conditions and investigate conditions with high mortality. Most critically ill patients are unable to comprehend or communicate and Substitute Decision Makers (SDMs) typically provide consent for their research participation. SDMs of critically ill patients may be overwhelmed by the patient's circumstances and the amount of medical information presented to them. Preliminary data suggest that SDMs prefer physician involvement in the consent process.

Primary Objective: To demonstrate the ability to implement a randomized controlled trial (RCT) evaluating two different approaches for introducing research coordinators (RC) to SDMs (physician introduction vs. non physician introduction) for participating in ICU research studies.

Secondary Objectives: To describe, among SDMs approached for consent to participate in an ICU research study by either physician or non-physician introduction (e.g., nurse, social worker)]: (a) the proportion of SDMs providing and declining consent, (b) the time between meeting eligibility criteria and sentinel events (being approached for consent, and either providing or declining consent), (c) reasons for SDMs providing or declining consent, and (d) agreement between questionnaires completed by SDMs and RCs and physicians regarding their acceptance of and comfort and satisfaction with the approach utilized.

Study Overview: We will conduct a multicentre pilot RCT of different methods (physician vs. non-physician introduction of research personnel) for approaching SDMs for consent for a loved one to participate in critical care research at 3 ICUs in Ontario.

Study Population: This study will focus on the approach to SDMs (n=99) of critically ill adults who are eligible (meet all inclusion criteria and have no exclusion criteria) to participate in a critical care research study in progress during the data collection period, and which requires SDM consent.

Interventions: In the intervention arm physicians will introduce RCs and study participation to SDMs using a standardized script. In the control arm RCs will either introduce themselves or be introduced by a non-physician member of the health care teams. RCs will complete an "Event Form" each time a critically ill adult is eligible to participate in a study. "Site Forms" and "Study Forms" will capture ICU-related information and studies in operation over the study period, respectively. We will administer 3 to 8 item questionnaires to SDMs, RCs and physicians involved in consent encounters to describe their acceptance of and comfort and satisfaction with the approach utilized.

Study Outcomes: To demonstrate the feasibility of an RCT evaluating 2 methods of approaching SDMs for consent for research participation. Feasibility will be defined as (i) ≤ 15% of physician introductions will be missed due to lack of physician availability (physician introduction arm) and (ii) cross-overs (from either arm to the other) will occur in ≤ 15% of encounters. We will demonstrate that ≤ 20% of introductions (following randomization) will be missed due to inability of the research team to contact an identified SDM and at least 70% and 50% of initial and subsequent SDM questionnaires will be returned.

Relevance: The Approach Study will provide valuable information for stakeholders committed to ensuring the ethical basis of critical care research; and will guide the design of a larger RCT examining how to best approach SDMs of critically ill patients. Moreover it will provide insight on how to best approach SDMs to make encounters more comfortable, credible, informed and less burdensome for them. The Approach Study will provide the framework for a larger phase 3 study examining how to best approach SDMs.

ELIGIBILITY:
Inclusion Criteria:

* SDMs of critically ill adults who are eligible (meet all inclusion criteria and have no exclusion criteria) to participate in a critical care research study in progress in the ICU

Exclusion Criteria:

* Eligible critically ill adults who die or are transferred out of a participating ICU prior to being screened by a RC
* Critically ill adults capable of providing primary consent for research participation.
* We will limit participation to initial encounters (the same patient will not be included more than once)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcome | 7 days
  Feasibility of the pilot study will be assessed by the following:
  1. We expect that (i) ≤ 15% of physician introductions will be missed due to lack of physician availability (physician introduction arm) and (ii) cross-overs (from either arm to the other) will occur in ≤ 15% on introductions.
  2. Following randomization, we expect that ≤ 20% of introductions will be missed due to inability of the RC to contact existing SDMs once identified (either intervention or control arm).
  3. We will obtain at least 70% of initial SDM questionnaires Part A and at least 50% of questionnaires Part B.

SECONDARY OUTCOMES:
Consent Obtained Vs Consent Declined | 7 days
  1. describe the proportion of SDMs providing and declining consent when approached by a RC or accompanied by the most responsible physician and when an update accompanies an introduction.
  2. determine the time interval between critically ill patients' meeting eligibility criteria and sentinel events.
  3. elucidate reasons why SDMs provide or decline consent
  4. assess agreement between SDMs, RCs and attending physicians acceptance of and comfort and satisfaction with the alternative approaches

CONTACTS AND LOCATIONS:
Overall Officials: Karen EA Burns, MD, FRCPC, MSc (Epid), Principal Investigator — St. Michael's Hospital, Toronto and the Keenan Research Centre/Li Ka Shing Knowledge Institute (Toronto)
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Sandham JD, Hull RD, Brant RF, Knox L, Pineo GF, Doig CJ, Laporta DP, Viner S, Passerini L, Devitt H, Kirby A, Jacka M; Canadian Critical Care Clinical Trials Group. A randomized, controlled trial of the use of pulmonary-artery catheters in high-risk surgical patients. N Engl J Med. 2003 Jan 2;348(1):5-14. doi: 10.1056/NEJMoa021108. PMID 12510037
- [Background] Cook D, Guyatt G, Marshall J, Leasa D, Fuller H, Hall R, Peters S, Rutledge F, Griffith L, McLellan A, Wood G, Kirby A. A comparison of sucralfate and ranitidine for the prevention of upper gastrointestinal bleeding in patients requiring mechanical ventilation. Canadian Critical Care Trials Group. N Engl J Med. 1998 Mar 19;338(12):791-7. doi: 10.1056/NEJM199803193381203. PMID 9504939
- [Background] SHIMKIN MB. The problem of experimentation on human beings. I. The research worker's point of view. Science. 1953 Feb 27;117(3035):205-7. doi: 10.1126/science.117.3035.205. No abstract available. PMID 13038475
- [Background] Coppolino M, Ackerson L. Do surrogate decision makers provide accurate consent for intensive care research? Chest. 2001 Feb;119(2):603-12. doi: 10.1378/chest.119.2.603. PMID 11171743
- [Background] Azoulay E, Chevret S, Leleu G, Pochard F, Barboteu M, Adrie C, Canoui P, Le Gall JR, Schlemmer B. Half the families of intensive care unit patients experience inadequate communication with physicians. Crit Care Med. 2000 Aug;28(8):3044-9. doi: 10.1097/00003246-200008000-00061. PMID 10966293
- [Background] Pochard F, Azoulay E, Chevret S, Lemaire F, Hubert P, Canoui P, Grassin M, Zittoun R, le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Symptoms of anxiety and depression in family members of intensive care unit patients: ethical hypothesis regarding decision-making capacity. Crit Care Med. 2001 Oct;29(10):1893-7. doi: 10.1097/00003246-200110000-00007. PMID 11588447
- [Background] Bolmsjo I, Hermeren G. Interviews with patients, family, and caregivers in amyotrophic lateral sclerosis: comparing needs. J Palliat Care. 2001 Winter;17(4):236-40. PMID 11813340
- [Background] Upadya A, Muralidharan V, Thorevska N, Amoateng-Adjepong Y, Manthous CA. Patient, physician, and family member understanding of living wills. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1430-5. doi: 10.1164/rccm.200206-503OC. Epub 2002 Sep 11. PMID 12406822
- [Background] Shalowitz DI, Garrett-Mayer E, Wendler D. The accuracy of surrogate decision makers: a systematic review. Arch Intern Med. 2006 Mar 13;166(5):493-7. doi: 10.1001/archinte.166.5.493. PMID 16534034
- [Background] Ciroldi M, Cariou A, Adrie C, Annane D, Castelain V, Cohen Y, Delahaye A, Joly LM, Galliot R, Garrouste-Orgeas M, Papazian L, Michel F, Barnes NK, Schlemmer B, Pochard F, Azoulay E. Ability of family members to predict patient's consent to critical care research. Intensive Care Med. 2007 May;33(5):807-813. doi: 10.1007/s00134-007-0582-6. Epub 2007 Mar 15. PMID 17361388
- [Background] Morley CJ, Lau R, Davis PG, Morse C. What do parents think about enrolling their premature babies in several research studies? Arch Dis Child Fetal Neonatal Ed. 2005 May;90(3):F225-8. doi: 10.1136/adc.2004.061986. PMID 15846012
- [Background] Scales DC, Smith OM, Pinto R, Barrett KA, Friedrich JO, Lazar NM, Cook DJ, Ferguson ND. Patients' preferences for enrolment into critical-care trials. Intensive Care Med. 2009 Oct;35(10):1703-12. doi: 10.1007/s00134-009-1552-y. Epub 2009 Jun 24. PMID 19551372
- [Background] Chenaud C, Merlani P, Verdon M, Ricou B. Who should consent for research in adult intensive care? Preferences of patients and their relatives: a pilot study. J Med Ethics. 2009 Nov;35(11):709-12. doi: 10.1136/jme.2008.028068. PMID 19880710
- [Background] Heyland DK, Rocker GM, Dodek PM, Kutsogiannis DJ, Konopad E, Cook DJ, Peters S, Tranmer JE, O'Callaghan CJ. Family satisfaction with care in the intensive care unit: results of a multiple center study. Crit Care Med. 2002 Jul;30(7):1413-8. doi: 10.1097/00003246-200207000-00002. PMID 12130954
- [Derived] Burns KE, Rizvi L, Smith OM, Lee Y, Lee J, Wang M, Brown M, Parker M, Premji A, Leung D, Hammond Mobilio M, Gotlib-Conn L, Nisenbaum R, Santos M, Li Y, Mehta S. Is there a role for physician involvement in introducing research to surrogate decision makers in the intensive care unit? (The Approach trial: a pilot mixed methods study). Intensive Care Med. 2015 Jan;41(1):58-67. doi: 10.1007/s00134-014-3558-3. Epub 2014 Dec 10. PMID 25491659